CLINICAL TRIAL: NCT06180889
Title: An Open, Randomized, Active-comparator-controlled, Multicenter Study to Assess the Efficacy and Safety of Different Doses of KN060 for the Prevention of Venous Thromboembolism in Patients Undergoing Unilateral Total Knee Arthroplasty.
Brief Title: Factor XI inhibiTion for the Prevention of Venous Thromboembolism in Patients Undergoing Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KN060-A-201
Record Dates: First submitted 2023-12-03; First posted 2023-12-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-12

CONDITIONS: Knee Arthroplasty, Total
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Enoxaparin (Active Comparator): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received enoxaparin for at least 10 days post-surgery.
  Interventions: Drug: Enoxaparin
- KN060 Low (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received KN060 low dose once post-surgery.
  Interventions: Drug: KN060 Low
- KN060 Middle (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received KN060 middle dose once post-surgery.
  Interventions: Drug: KN060 Middle
- KN060 Hight (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received KN060 hight dose once post-surgery.
  Interventions: Drug: KN060 Hight

INTERVENTIONS:
Drug: Enoxaparin — 40 mg enoxaparin administered as subcutaneous injection once daily
  Arms: Enoxaparin
Drug: KN060 Low — Single dose of KN060 administered as intravenous infusion
  Arms: KN060 Low (post-surgery)
Drug: KN060 Middle — Single dose of KN060 administered as intravenous infusion
  Arms: KN060 Middle (post-surgery)
Drug: KN060 Hight — Single dose of KN060 administered as intravenous infusion
  Arms: KN060 Hight (post-surgery)

SUMMARY:
This study was to compare the study drug KN060 to enoxaparin, for the prevention of blood clotting and safety in patients undergoing total knee arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 75 years old (including the cut-off value);
2. undergoing unilateral Total Knee Arthroplasty (TKA);
3. Voluntarily participate in the study and sign a written informed consent;

Exclusion Criteria:

1. There is a high risk of bleeding or abnormal bleeding related indicators:
2. Evidence of venous thrombosis, such as the presence of related symptoms or auxiliary tests indicating thrombosis; Or have a history of venous embolic disease.
3. Acute myocardial infarction or ischemic stroke occurred within 6 months before screening.
4. Presence of malignant tumors or history of malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite endpoint consisting of asymptomatic DVT as detected by mandatory bilateral venography, objectively confirmed symptomatic DVT, non-fatal PE, fatal PE, unexplained death for which PE cannot be excluded | Up to 14 days
  DVT - Deep vein thrombosis / PE - Pulmonary embolism. All suspected events were reviewed and classified by the investigator

SECONDARY OUTCOMES:
Incidence of composite endpoint of major and clinically relevant non-major bleeding | Up to 14 days
  All suspected events were reviewed and classified by the investigator
Incidence of composite endpoint consisting of asymptomatic DVT as detected by mandatory bilateral venography, objectively confirmed symptomatic DVT, non-fatal PE, fatal PE, unexplained death for which PE cannot be excluded | Up to 35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of symptomatic DVT, non-fatal PE | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of fatal PE | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of unexplained death for which PE cannot be excluded | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of composite endpoint of major and clinically relevant non-major bleeding | Up to 35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of bleeding | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of major bleeding | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of clinically relevant non-major bleeding | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Incidence of treatment emergent adverse event/adverse drug reaction | Up to 14 \35\100 days
  All suspected events were reviewed and classified by the investigator
Plasma Concentration of KN060 | Up to 100 days
Pharmacodynamics index: Changes of plasma concentration of Free FⅪ from baseline; | Up to 100 days
  Free FⅪ: Free Factor XI; Factor XI is a clotting factor.
Pharmacodynamics index: Changes of FⅪ activity from baseline; | Up to 100 days
  FⅪ: Factor XI; Factor XI is a clotting factor.
Pharmacodynamics index: Changes of APTT from baseline; | Up to 100 days
  APTT: activated partial thromboplastin time;

CONTACTS AND LOCATIONS:
Overall Officials: Xianlong Zhang, Doctor, Principal Investigator — Shanghai 6th People's Hospital; Feng Yin, Doctor, Principal Investigator — Shanghai East Hospital of Tongji University; Zhenjun Yao, Doctor, Principal Investigator — Fudan University; Shijun Gao, Doctor, Principal Investigator — Hebei Medical University Third Hospital; Jun Lu, Doctor, Principal Investigator — Zhongda Hospital; Xinshe Zhou, Doctor, Principal Investigator — The First Affiliated Hospital Of Bengbu Medicai College; Rende Ning, Doctor, Principal Investigator — Hefei First People's Hospital; Lidong Wu, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Wenming Zhang, Doctor, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Yayi Xia, Doctor, Principal Investigator — Lanzhou University Second Hospital; Song Chen, Doctor, Principal Investigator — The Third Hospital of Changsha; Tan Lu, Doctor, Principal Investigator — The First Affiliated Hospital Of Xingxiang Medical University; Chunming Huang, Doctor, Principal Investigator — The People's Hospital of Gaozhou; Jun Xiao, Doctor, Principal Investigator — Tongji Hospital; Pengde Kang, Doctor, Principal Investigator — West China Hospital; Min Dai, Doctor, Principal Investigator — The First Affiliated Hospital of Nanchang University; Wei Huang, Doctor, Principal Investigator — First Affiliated Hospital of Chongqing Medical University; Jiangwei Li, Doctor, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University; Bensen Tang, Doctor, Principal Investigator — Beijing Jishuitan Hosptial Guizhou Hospital; Li Sun, Doctor, Principal Investigator — Guizhou Provincial Peoples Hospital; Xu Cai, Doctor, Principal Investigator — Beijing Tsinghua Changgeng Hospital; Xin Wang, Doctor, Principal Investigator — Yantai Yuhuangding Hospital; Huiwu Li, Doctor, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No